CLINICAL TRIAL: NCT04365868
Title: A Seamless, Adaptive, Phase 2b/3, Double-Blind, Randomized, Placebo-controlled, Multicenter, International Study Evaluating the Efficacy and Safety of Belapectin (GR MD-02) for the Prevention of Esophageal Varices in NASH Cirrhosis
Brief Title: Study Evaluating the Efficacy and Safety of Belapectin for the Prevention of Esophageal Varices in NASH Cirrhosis
Acronym: NAVIGATE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Based on FDA feedback, Stage 1 of NAVIGATE was analyzed as a stand-alone trial. Study was not prematurely terminated for safety reasons.
Sponsor: Galectin Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GT-031
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Prevention of Esophageal Varices; NASH - Nonalcoholic Steatohepatitis; Cirrhosis
Keywords: esophageal varices; belapectin; GR-MD-02; portal hypertension; nonalcoholic steatohepatitis (NASH) cirrhosis; NASH; cirrhosis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis; Esophageal and Gastric Varices; Hypertension, Portal | interventions — belapectin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- belapectin 2 mg/kg lean body mass (LBM) (Experimental): Phase 2b: Belapectin 2 mg/kg lean body mass administered intravenously (IV) every other week for 78 weeks (18 months)
  Phase 3: The patient will be switched to the optimal dose
  Interventions: Drug: belapectin
- belapectin 4 mg/kg lean body mass (LBM) (Experimental): Phase 2b: Belapectin 4 mg/kg lean body mass administered intravenously (IV) every other week for 78 weeks (18 months)
  Phase 3: The patient will be switched to the optimal dose
  Interventions: Drug: belapectin
- Placebo (Placebo Comparator): Phase 2b: Placebo, administered intravenously (IV) every other week for 78 weeks (18 months)
  Phase 3:Placebo, administered intravenously (IV) every other week for 78 weeks (18 months)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: belapectin — intravenous
  Other Names: GR-MD-02; galactoarabino rhamnogalacturonate
  Arms: belapectin 2 mg/kg lean body mass (LBM); belapectin 4 mg/kg lean body mass (LBM)
Drug: Placebo — intravenous
  Arms: Placebo

SUMMARY:
This seamless, adaptive, two-stage, Phase 2b/3, randomized, double-blind, multicenter, parallel-groups, placebo-controlled study will assess the efficacy, safety, and tolerability of belapectin compared with placebo in patients with nonalcoholic steatohepatitis (NASH) cirrhosis and clinical signs of portal hypertension but without esophageal varices at baseline.

ELIGIBILITY:
Inclusion Criteria:

Each subject must meet all of the following criteria to be enrolled in this study:

1. Is male or female, ≥ 18 and ≤ 75 years of age at the time of Screening.
2. Is willing and able to provide written informed consent prior to the initiation of any study-specific procedures.
3. Has evidence of portal hypertension, with either one of the following:

   1. platelet count <150,000/mm3

      OR
   2. documented hepatic venous pressure gradient (HVPG) measurement >6 mmHg

      OR
   3. at least two of the following:

      * spleen size ≥14 cm (documented by ultrasound, MRI, or CT scan)
      * abdominal collateral circulation (documented by ultrasound, MRI, or CT scan or physical examination, ie, caput medusae)
      * documented liver transient elastography (eg, FibroScan) ≥20 kilopascals (kPa).
      * aspartate aminotransferase (AST)/alanine aminotransferase (ALT) >1.
4. Has a history confirming nonalcoholic steatohepatitis (NASH) cirrhosis, with at least one of the following:

   * There is a historical liver biopsy showing cirrhosis with steatohepatitis. There is no evidence for a competing etiology for the cirrhosis.
   * There is a historical liver biopsy showing steatohepatitis, and there is evidence of cirrhosis from clinical or imaging data or a second liver biopsy showing cirrhosis without all features of NASH (as the histological NASH lesions may have burnt out). There is no evidence for a competing etiology. There is at least 1 co-existing metabolic comorbidity at Screening: obesity (with either body mass index [BMI] ≥30 kg/m2 or waist circumference ≥102 cm [40 in, men] or ≥88 cm [35 in, women], or by ethnically appropriate cutpoints); hypertension (either on anti hypertensive drug therapy for at least 1 year or systolic/diastolic blood pressure (BP) >140/80 mm Hg); Type 2 diabetes (glycated hemoglobin [HbA1c] ≥6.5%, or on anti-diabetic medication for at least 1 year); or dyslipidemia (triglycerides ≥150 mg/dL or on drug therapy for hypertriglyceridemia for at least 6 months; high-density lipoprotein cholesterol ≤40 mg/dL [men] or ≤50 mg/dL [women]) to corroborate a diagnosis of nonalcoholic fatty liver disease (NAFLD).
   * There is a historical liver biopsy showing cirrhosis with steatosis but not steatohepatitis. There is no evidence for a competing etiology. There are at least 2 co-existing (or history of) metabolic comorbidities (with obesity or diabetes being one of them) to corroborate a diagnosis of NAFLD.
   * There is a historical liver biopsy showing steatosis but now with cirrhosis either by clinical examination, imaging, or biopsy. If there is a current biopsy, it does not show evidence of steatosis or steatohepatitis as histological lesions may have burned out. There is no evidence for a competing etiology. There are at least 2 co existing (or history of) metabolic comorbidities (with obesity or diabetes being one of them) to corroborate a diagnosis of NAFLD.
   * Patient with cirrhosis with current or previous imaging showing steatosis. There is no liver histology available. There is no evidence for a competing etiology. There are at least two co-existing or history of metabolic comorbidities with obesity or diabetes being one of them to corroborate a diagnosis of NAFLD.
   * For patients not meeting the above mentioned criteria, a screening liver biopsy is necessary.

   Note: All liver biopsy blocks and/or slides for eligibility assessments (including those from historical biopsies) will be reviewed by the central study pathologist while the subject is in Screening. Results from the central study pathologist must be available before the subject is randomized.
5. Absence of hepatocellular carcinoma (HCC) by valid imaging (eg, ultrasound, CT scan, or MRI) within 6 months prior to randomization. If no such imaging result is available, then ultrasound imaging should be performed as part of standard of care.
6. Patients with diabetes mellitus can be enrolled, if they are adequately controlled on a stable dose or doses of antidiabetic medication(s) for at least 3 months before Screening, and their screening HbA1c is ≤9.5%.
7. Patients on vitamin E or pioglitazone can be enrolled if they are on a stable dose and regimen for at least 3 months before screening, and the dose is expected to be held constant during the trial.
8. Patients on a statin can be enrolled if they are on a stable regimen for at least 3 months before Screening, and expected to be held stable during the trial.
9. Is not pregnant and must have a negative serum pregnancy test result prior to randomization.
10. Is of non-childbearing potential or if a fertile man or woman participating in heterosexual relations, agrees to use two acceptable means of contraception (ie, 2 effective methods of contraception, one of which must be a physical barrier method [eg, male or female condom, diaphragm] when combined with a highly effective method of contraception [ie, a method with a failure rate of <1% per year when used consistently and correctly]) throughout his/her participation in this study and for 90 days after discontinuation of study treatment.

    Highly effective forms of contraception include:
    * combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (such as oral, intravaginal, transdermal) methods
    * progestogen-only hormonal contraception associated with inhibition of ovulation (such as oral, injectable, implantable)
    * hormone-releasing intrauterine system (IUS)
    * intrauterine device (IUD)
    * bilateral tubal occlusion
    * a vasectomized partner, provided that partner is the sole sexual partner of the women of childbearing potential trial participant and that the vasectomized partner has received medical assessment of the surgical success
    * sexual abstinence (ie, a refraining from heterosexual intercourse during the entire period of the clinical trial, if it is the preferred and usual lifestyle of the subject).

    Surgically sterile males and females are not required to use contraception provided they have been considered surgically sterile for at least 6 months. Surgical sterility includes history of surgically successful vasectomy, hysterectomy, or bilateral salpingo-oophorectomy. Postmenopausal women who have been amenorrheic for at least 2 years at the time of Screening will be considered sterile.
11. If a lactating woman, agrees to discontinue nursing before the start of study treatment and refrain from nursing until 90 days after the last dose of study treatment.
12. If a man, agrees to refrain from sperm donation throughout the study period and for a period of 90 days following the last dose of investigational medicinal product (IMP). Female subjects may not begin a cycle of ova donation or harvest throughout the study period and for a period of 90 days following the last dose of IMP.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from the study:

1. Presence of esophageal, gastroesophageal, or isolated gastric varices, based on an upper gastrointestinal (GI) esophagogastroduodenoscopy (EGD) exam conducted during Screening. Patients with portal hypertensive gastropathy could be enrolled.
2. History of hepatic cirrhosis decompensation including any episode of variceal bleeding, ascites not controlled by medication, spontaneous bacterial peritonitis or overt hepatic encephalopathy (West Haven grade ≥2 as assessed by the principal investigator), OR develops signs of hepatic cirrhosis decompensation during Screening.
3. Known or suspected abuse of alcohol (>20 g/day for women or >30 g/day for men [on average per day]), as per medical history. Significant alcohol consumption is defined as more than 20 grams per day in females and more than 30 grams per day in males. On average, a standard drink in the United States is considered to be 14 grams of alcohol, equivalent to 12 fluid ounces of regular beer (5% alcohol), 5 fluid ounces of table wine (12% alcohol), or 1.5 fluid ounces of 80 proof spirits (40% alcohol).
4. Alcohol dependence (ie, a score >8 on the Alcohol Use Disorders Identification Test)
5. Narcotics or any other drug abuse or dependence in the last 5 years
6. Prior trans-jugular intrahepatic portal-systemic (TIPS) shunt procedure
7. Documented causes of liver disease other than NASH, including but not restricted to:

   * Viral hepatitis, unless eradicated at least 3 years prior to Screening

     * acute hepatitis A infection (presence of hepatitis A immunoglobulin M [IgM] at Screening)
     * positive hepatitis B surface antigen
     * positive hepatitis C virus (HCV) ribonucleic acid (to be performed prior to randomization in case of positive HCV antibody)
   * Documented drug-induced liver disease
   * Alcoholic liver disease
   * Autoimmune hepatitis
   * Wilson's disease
   * Hemochromatosis
   * Primary biliary cholangitis
   * Primary sclerosing cholangitis
   * Genetic hemochromatosis
   * History or planned liver transplantation
   * Alpha-1 antitrypsin deficiency
8. History of human immunodeficiency virus (HIV), or positive HIV test at Screening
9. Any of the following test or score:

   * serum alanine aminotransferase (ALT) > 5 × upper limit of normal (ULN)*
   * serum aspartate aminotransferase (AST) > 5 × ULN*

     *Screening values will be obtained at Screening Visit 1 (SV1) and Screening Visit 2(SV2) (which will be separated by 2 to 4 weeks). A second screening value that is >50% higher than the first value should prompt re-evaluation of the severity of the underlying liver disease and eligibility for this trial. If a transaminase level at SV2 is >33% different from the level at SV1, then additional measurements should be performed at Screening Visit 3 (SV3). In such cases, the baseline transaminase levels will be established for subjects using the mean value of 4 evaluations [ie, at SV1, SV2, SV3, and Baseline (ie, pre-dose during Visit 1)].
   * serum alkaline phosphatase (ALP) > 2 × ULN
   * mean platelet count < 50,000/mm3
   * total bilirubin ≥ 2.0 mg/dL (subjects with a documented history of Gilbert's syndrome can be enrolled if the direct bilirubin is within normal reference range)
   * model for end-stage liver disease (MELD) score ≥12
   * Child-Turcotte-Pugh (CTP) Score ≥7 Note: Following Phase 2b, subjects with CTP scores ≥7 may be enrolled if recommended* by the Data Safety Monitoring Board (DSMB) and approved by the Trial Steering Committee (TSC), based on the planned interim analysis (IA). [*based on DSMB review of preliminary results from a separate hepatic impairment clinical trial (Study GT-032) which is assessing belapectin safety and pharmacokinetic (PK) in cirrhotic subjects with CTP scores ≥7.
   * estimated glomerular filtration rate < 45 mL/min* *Note: per Modification of Diet in Renal Disease algorithm
10. Taking an angiotensin converting enzyme inhibitor, angiotensin II receptor blocker, or β-1 selective adrenergic receptor inhibitor, unless on a stable regimen for at least 3 months prior to Screening and no changes in the regimen are anticipated during the study. Subjects taking a non-selective beta blocker are not eligible to be enrolled (Investigators are encouraged to substitute another medication, if clinically warranted).
11. History of major surgery during Screening.
12. History of a solid organ transplant requiring immunosuppressive therapy.
13. History of bariatric surgery within 1 year of randomization, or plan to undergo bariatric surgery during the study.
14. Has positive screening test for illicit drugs of abuse at Screening.
15. Has participated in an investigational new drug study within 30 days or 5 half-lives whichever is longer, prior to randomization.
16. Has a history of malignancy within 5 years of randomization, except for basal cell carcinoma, squamous cell carcinoma, and adequately treated in situ uterine cervical cancer.
17. Has clinically significant cardiovascular disease (eg, uncontrolled hypertension, myocardial infarction, unstable angina), New York Heart Association Grade II or greater congestive heart failure, serious cardiac arrhythmia requiring intervention (eg, pacemaker/ablation) or Grade II or greater peripheral vascular disease.
18. Has a history of clinically significant hematologic, renal, hepatic, pulmonary, neurological, psychiatric, gastrointestinal, systemic inflammatory, metabolic or endocrine disorder or any other condition that, in the opinion of the Investigator, renders the subject a poor candidate for inclusion into the study.
19. Has known allergies to the IMP or any of its excipients.
20. Has previously received belapectin within 6 months of randomization.
21. Is an employee or family member of the Investigator or study center personnel.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-04-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in the belapectin treatment groups who develop new esophageal varices at 78 weeks [18 months] of treatment compared to placebo | At 78 weeks [18 months]
  Proportion of patients in the belapectin treatment groups who develop new esophageal varices at 78 weeks [18 months] of treatment compared to placebo

SECONDARY OUTCOMES:
Efficacy: Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop varices (esophageal or gastric) requiring treatment | Through study end, 78 weeks or 156 weeks
  Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop varices (esophageal or gastric) requiring treatment
Efficacy: Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop variceal bleed requiring hospitalization | Through study end, 78 weeks or 156 weeks
  Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop variceal bleed requiring hospitalization
Efficacy: Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop clinically significant ascites requiring hospitalization | Through study end, 78 weeks or 156 weeks
  Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop clinically significant ascites requiring hospitalization
Efficacy: Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop spontaneous bacterial peritonitis | Through study end, 78 weeks or 156 weeks
  Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop spontaneous bacterial peritonitis
Efficacy: Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop hepatic encephalopathy (West Haven score ≥2 and requiring hospitalization) | Through study end, 78 weeks or 156 weeks
  Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop hepatic encephalopathy (West Haven score ≥2 and requiring hospitalization)
Efficacy: Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop mortality (all-cause) | Through study end, 78 weeks or 156 weeks
  Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop mortality (all-cause)
Efficacy: Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop liver transplant | Through study end, 78 weeks or 156 weeks
  Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop liver transplant
Efficacy: Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop model for end-stage liver disease (MELD) score ≥15 | Through study end, 78 weeks or 156 weeks
  Cumulative incidence rate of patients in the belapectin treatment groups, compared to placebo, who develop model for end-stage liver disease (MELD) score ≥15
Efficacy: Cumulative incidence rate of patients in the belapectin Phase 3 treatment group who progress to large varices (gastric or esophageal) or develop red wales compared to placebo. | Through study end, 78 weeks or 156 weeks
  Cumulative incidence rate of patients in the belapectin Phase 3 treatment group who progress to large varices (gastric or esophageal) or develop red wales compared to placebo
Efficacy: Event-free survival by time to first cirrhosis related clinical event, progression to large varices or red wales | Through study end, 78 weeks or 156 weeks
  Event-free survival by time to first cirrhosis related clinical event, progression to large varices or red wales
Efficacy: Event-free survival by time to first cirrhosis related clinical event, esophageal variceal hemorrhage requiring hospitalization | Through study end, 78 weeks or 156 weeks
  Event-free survival by time to first cirrhosis related clinical event, esophageal variceal hemorrhage requiring hospitalization
Efficacy: Event-free survival by time to first cirrhosis related clinical event, clinically significant ascites requiring hospitalization | Through study end, 78 weeks or 156 weeks
  Event-free survival by time to first cirrhosis related clinical event, clinically significant ascites requiring hospitalization
Efficacy: Event-free survival by time to first cirrhosis related clinical event, spontaneous bacterial peritonitis | Through study end, 78 weeks or 156 weeks
  Event-free survival by time to first cirrhosis related clinical event, spontaneous bacterial peritonitis
Efficacy: Event-free survival by time to first cirrhosis related clinical event, overt hepatic encephalopathy (West Haven score ≥2 and requiring hospitalization) | Through study end, 78 weeks or 156 weeks
  Event-free survival by time to first cirrhosis related clinical event, overt hepatic encephalopathy (West Haven score ≥2 and requiring hospitalization)
Efficacy: Event-free survival by time to first cirrhosis related clinical event, Child-Turcotte-Pugh (CTP) score increase of ≥2 points (from baseline) | Through study end, 78 weeks or 156 weeks
  Event-free survival by time to first cirrhosis related clinical event, Child-Turcotte-Pugh (CTP) score increase of ≥2 points (from baseline)
Efficacy: Event-free survival by time to first cirrhosis related clinical event, model for end-stage liver disease (MELD) score increase to ≥15 as measured on 2 consecutive occasions | Through study end, 78 weeks or 156 weeks
  Event-free survival by time to first cirrhosis related clinical event, model for end-stage liver disease (MELD) score increase to ≥15 as measured on 2 consecutive occasions
Efficacy: Event-free survival by time to first cirrhosis related clinical event, liver transplant | Through study end, 78 weeks or 156 weeks
  Event-free survival by time to first cirrhosis related clinical event, liver transplant
Efficacy: Event-free survival by time to first cirrhosis related clinical event, liver-related death | Through study end, 78 weeks or 156 weeks
  Event-free survival by time to first cirrhosis related clinical event, liver-related death

OTHER OUTCOMES:
Exploratory Efficacy:Change in liver stiffness measurement (LSM), baseline-adjusted, as determined by vibration controlled transient elastography (VCTE) (FibroScan) exams during Phase 2b and Phase 3 | Through study end, 78 weeks or 156 weeks
  Change in liver stiffness measurement (LSM), baseline-adjusted, as determined by vibration controlled transient elastography (VCTE) (FibroScan) exams during Phase 2b and Phase 3
Exploratory Efficacy: Difference in Chronic Liver Disease Questionnaire (CLDQ) scores between belapectin and placebo treatment during Phase 2b and Phase 3 | Through study end, 78 weeks or 156 weeks
  The difference in Chronic Liver Disease Questionnaire scores between belapectin and placebo treatment during Phase 2b and Phase 3 will be observed; Subject responses to the questionnaire are based on a scale from 1 to 7, with 1 being maximum frequency and 7 being none at all. Scores indicative of higher frequency, indicate worse outcomes.
Safety: Incidence of adverse events | Through study end, 78 weeks or 156 weeks
  Incidence of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Khurram Jamil, M.D., Study Director — Galectin Therapeutics Inc.
Locations (156):
- United States (81):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Digestive Health Specialists, Dothan, Alabama
  - The Institute for Liver Health, Chandler, Arizona
  - Arizona Liver Health - Glendale, Glendale, Arizona
  - Institute for Liver Health - Tucson, Tucson, Arizona
  - Liver Wellness Center - Little Rock, Little Rock, Arkansas
  - Hope Clinical Research, Inc., Canoga Park, California
  - Southern California GI & Liver Centers, Coronado, California
  - University of California San Diego Medical Center -La Jolla Multi-Specialty Clinics- Perlman Offices, La Jolla, California
  - Om Research LLC, Lancaster, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - inSite Digestive Health Care - Orange, Orange, California
  - California Liver Research Institute, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Integrity Clinical Research, LLC (ICR SITES) - Doral, Doral, Florida
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - Mayo Clinic Hospital - Florida, Jacksonville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - ClinCloud LLC, Maitland, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Genoma Research Group, Inc., Miami, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Guardian Angel Health Services, Inc., Tampa, Florida
  - Florida Medical Center & Research, Zephyrhills, Florida
  - Digestive Healthcare of Georgia, P.C., Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, LLC, Macon, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Loyola University Health System, Maywood, Illinois
  - IU Health University Hospital, Indianapolis, Indiana
  - Michiana Gastroenterology, Inc., South Bend, Indiana
  - Kansas Medical Clinic PA, Topeka, Kansas
  - University of Louisville Physicians - Cardiovascular Medicine Physicians Outpatient Center, Louisville, Kentucky
  - Tandem Clinical Research, LLC, Marrero, Louisiana
  - Tulane Cancer Center, New Orleans, Louisiana
  - Mercy Medical Center - The Institute for Digestive Health and Liver Disease, Baltimore, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System - Hemophilia and Thrombosis Treatment Center, Detroit, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - Southern Therapy and Advanced Research (STAR) - Jackson, Jackson, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Excel Clinical Research - Las Vegas, Las Vegas, Nevada
  - Mount Sinai Beth Israel, New York, New York
  - NYU Langone Medical Center, New York, New York
  - NewYork-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - UNC-Chapel Hill School of Medicine, Chapel Hill, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Lucas Research, Morehead City, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - University of Cincinnati Physicians Company, LLC, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Jefferson Digestive Health Institute - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC) - The Center for Liver Diseases, Pittsburgh, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Galen Medical Group - Ziegler Plaza, Chattanooga, Tennessee
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - Gastro One - GI Diagnostic and Therapeutic Endoscopy Center - 1310 Wolf Park, Germantown, Tennessee
  - Associates in Gastroenterology, Hermitage, Tennessee
  - East Tennessee Research Institute - Gastrointestinal Associates of Northeast Tennessee, P.C., Johnson City, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Liver Specialists of Texas, Austin, Texas
  - Methodist Transplant Physicians, Dallas, Texas
  - Texoma Liver Center PLLC. - Denison, Denison, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Baylor College of Medicine - Baylor Clinic - Abdominal Transplant & Liver Disease Clinic, Houston, Texas
  - Pioneer Research Solutions Inc - Houston - Stancliff Rd, Houston, Texas
  - The Texas Liver Institute, Inc., San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Impact Research Institute, Waco, Texas
  - University of Utah Health Care - UUHC - Kidney & Liver Clinic, Salt Lake City, Utah
  - University of Virginia School of Medicine, Charlottesville, Virginia
  - Gastroenterology Associates of Fredericksburg, Fredericksburg, Virginia
  - Bon Secours Liver Institute of Virginia - Newport News, Newport News, Virginia
  - Bon Secours Liver Institute of Virginia - Richmond, Richmond, Virginia
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
  - Velocity Clinical Research, Spokane, Spokane, Washington
- Argentina (3):
  - Hospital Italiano de Buenos Aires, Buenos Aires, ARG
  - Hospital Británico de Buenos Aires, Buenos Aires, ARG
  - Centro de Investigaciones Metabólicas (CINME), Capital Federal, ARG
- Australia (5):
  - Nepean Hospital, Kingswood, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre Clayton, Clayton, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (5):
  - Antwerp University Hospital, Edegem, Antwerpen
  - Clinique Universitaire De Bruxelles Hôpital Erasme VZW, Brussels, BEL
  - AZ Maria Middelares, Ghent, VOV
  - Universitair Ziekenhuis Gent, Ghent, VOV
  - Groupe sante CHC - Clinique du MontLegia, Liège, WLG
- Canada (5):
  - University of Calgary - Heritage Medical Research Clinic - Foothills Hospital Center, Calgary, Alberta
  - Pacific Gastroenterology Associates, Vancouver, British Columbia
  - Brampton Civic Hospital, Brampton, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
- Chile (4):
  - Hospital de La Serena, La Serena, CHL
  - Clínica Universidad de los Andes, Santiago, CHL
  - Centro de Investigaciones Clinicas Vina del Mar, Viña del Mar, CHL
  - Hospital Clínico Universidad de Chile, Santiago
- France (10):
  - Centre Hospitalier Universitaire d'Amiens, Amiens
  - Hôpital Avicenne, Bobigny
  - CHU Hôpital Henri Mondor, Créteil
  - CHU de Grenoble, Grenoble
  - Hôpital de la Croix-Rousse, Lyon
  - CHRU Montpellier - Saint Eloi, Montpellier
  - CHU Nancy - Hôpital Brabois, Nancy
  - CHU de Nice - L'Archet, Nice
  - Hôpital Cochin, Paris
  - Hôpitaux Universitaires de Strasbourg - Hôpital Civil, Strasbourg
- Germany (3):
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz, Mainz, Rhineland-Palatinate
  - EUGASTRO GmbH, Leipzig, Saxony
  - Goethe-Universität Frankfurt am Main, Frankfurt am Main
- Israel (8):
  - Soroka Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Hadassah Ein Karem Hospital, Jerusalem
  - Holy Family Hospital, Nazareth
  - Rabin Medical Center - Beilinson Hospital, Petah Tikva
  - The Chaim Sheba Medical Center - The Center for Liver Diseases, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Mexico (13):
  - CICPA Centro de Investigación Clinica del Pacifico, Acapulco de Juárez, Guerrero
  - Centro de Investigacion Medico Biologica y Terapia Avanzada SC, Guadalajara, Jalisco
  - Investigacion Biomedica para el desarrollo de farmacos SA de CV, Zapopan, Jalisco
  - Investigacion Biomedica para el desarrollo de farmacos SA de CV, Benito Juárez, Mexico City
  - CEMDEC SA de CV Centro Mexicano de Desarrollo de Estudios Clinicos, Cuauhtémoc, Mexico City
  - Centro Especializado en Diabetes, Obesidad y Pevencion de enfermedades Cadiovasculares SC., Miguel Hidalgo, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez Servicio de Gastroenterología, Monterrey, Nuevo León
  - Oaxaca Site Management Organization SC., Oaxaca City, Oaxaca
  - Consultorio Medico, Ciudad de Mexico, State of Mexico
  - Medical Care and Research SA de CV, Mérida, Yucatán
  - Centro de Investigación Medica de Aguascalientes, Aguascalientes
  - MEDIVEST Centro de Investigacion integral, Chihuahua City
  - Centro de Investigacion Clinica de Oaxaca, Oaxaca City
- Poland (4):
  - SP CSK im Prof. Kornela Gibińskiego Śląskiego Uniwersytetu Medycznego w Katowicach, Katowice, Silesian Voivodeship
  - ID Clinic, Mysłowice, Silesian Voivodeship
  - Medyczny Katedra i Klinika Chorób Zakaźnych, Chorób Wątroby i Nabytych Niedoborów Odpornościowych, Wroclaw
  - Medical University of Lodz, Lodz, Łódź Voivodeship
- Fundacion de Investigacion de Diego, San Juan, Puerto Rico
- South Korea (4):
  - Hanyang University Seoul Hospital, Seoul, KOR
  - Yonsei University, Wonju Severance Christian Hospital, Seoul, KOR
  - Yonsei University, Wonju Severance Christian Hospital, Wŏnju, KOR
  - Digestive Research Alliance of Michiana, LLC, Incheon
- Spain (8):
  - Hospital Universitario 12 de Octubre, Madrid, ESP
  - Hospital del Mar Research Institute, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda
  - Complexo Hospitalario Universitario de Pontevedra, Pontevedra
  - Hospital Universitario Marqués de Valdecilla, Santander
  - Hospital Universitario Virgen del Rocío, Seville
- United Kingdom (2):
  - King's College Hospital NHS Foundation Trust, London, GBR
  - The University of Nottingham - Nottingham Digestive Diseases Centre Biomedical Research Unit, Nottingham, NGM

IPD SHARING:
Plan to Share IPD: No